CLINICAL TRIAL: NCT06688812
Title: Comparative Effects of Perceptual Motor Training and Repetitive Facilitation Exercises on Upper Limb Quality of Movement and Motor Function in Stroke Patients
Brief Title: Comparing Perceptual Motor Training and Repetitive Facilitation Exercises on UE in Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0253
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: exercise; motor skills; rehabilitation; stroke; upper extremity
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Perceptual Motor Training with Routine Physical Therapy (Experimental): Group A will receive treatment session of 60 minutes including Perceptual motor training for 40 minutes along with routine physical therapy of 20 minutes. Treatment session will be given 4 days per week for 8 weeks. Effects will be measured at baseline, 4th week and post intervention.
  Interventions: Other: Perceptual Motor Training
- Group B Repetitive Facilitation Exercises with Routine Physical Therapy (Experimental): Group B will receive treatment session of 60 minutes including Repetitive facilitation exercises for 40 minutes along with routine physical therapy of 20 minutes. Treatment session will be given 4 days per week for 8 weeks. Effects will be measured at baseline, 4th week and post intervention.
  Interventions: Other: Repetitive Facilitation Exercises

INTERVENTIONS:
Other: Perceptual Motor Training — 8 set of exercises
  1. Balance training and related exercises
  2. Tones of awareness training, body parts' role and related exercises
  3. Space awareness training and related exercises
  4. Perception of shape training and related exercises
  5. Visual perception training and related exercise.
  6. Kinesthetic-tactile perception training and related exercises
  7. Auditory perception training and related exercises
  8. Eye and hand coordination, ﬁne motor movements and related Exercises
  Arms: Group A Perceptual Motor Training with Routine Physical Therapy
Other: Repetitive Facilitation Exercises — Eight set of exercises:
  1. Shoulder Flexion with 90° Elbow Flexion (Supine).
  2. Shoulder Horizontal Extension/Flexion with Elbow flexion (supine).
  3. Complex Shoulder and Upper Limb Movements (Supine)
  4. Shoulder Flexion/Abduction/External Rotation with Elbow and Forearm Supination (Supine)
  5. Forearm Supination/Pronation with 90° Elbow Flexion (Sitting)
  6. Wrist Extension and Forearm Pronation with Finger Extension (Supine)
  7. Finger Extension with Wrist Flexion (Supine)
  8. Finger Extension/Flexion with Wrist Flexion (Sitting) • Therapist facilitate the movement by rubbing, tapping and gentle stretching.
  Arms: Group B Repetitive Facilitation Exercises with Routine Physical Therapy

SUMMARY:
The aim of the study is to determine the comparative effects of perceptual motor training and repetitive facilitation exercises on upper limb quality of movement and motor function in Stroke patients.

DETAILED DESCRIPTION:
Perceptual-motor training enhances proprioception, spatial awareness, and coordination through object manipulation. On the other hand, Repetitive facilitation exercises aim to improve motor control and reduce spasticity by stimulating muscles repetitively. Decreased dexterity, coordination, muscle tone abnormalities, and diminished sensation are frequently observed in stroke patients. Effective rehabilitation in daily tasks depends on coordinated efforts among muscles, joints, and body segments, influenced by environmental factors and personal constraints. Visual input, perception, and cognitive processing play crucial roles in action planning during rehabilitation.

This is a randomized clinical trial. The data will be collected from DHQ hospital, Sargodha. 50 stroke patients will be included using convenience sampling. The participants who meet the inclusion criteria will be randomly allocated into two groups. Twenty-five participants will be included in both Groups A and B. Group A (perceptual motor training with routine physical therapy) and Group B (Repetitive facilitation exercises with routine physical therapy) will receive 60 minutes treatment session that consists of 40 minutes of intervention and 20 minutes of routine physical therapy four sessions per week for 8 weeks.

Quality of movement will be assessed using Motor Evaluation Scale for Upper Extremity in Stroke Patients (MESUPES) and motor function by Fugl-Meyer Assessment (FMA-UE) Assessments will occur at baseline, 4 weeks, and 8 weeks. Data analysis will utilize SPSS version 27 for Windows, with statistical significance set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria;

* Both male and female patients.
* Age 40-65 years
* 1st ever stroke confirmed by MRI
* mild-to-moderate upper-limb motor paralysis
* sub-acute and chronic stroke patients
* ability to understand tasks such as evaluations in the intervention
* Modified Ashworth scale score < 3
* Mini Mental State Examination Score should be>24 out of 30

Exclusion Criteria:

* Participants who have a history of significant neurological or psychiatric disorders, other than stroke, that could interfere with upper limb motor recovery
* Patients with pain, contracture and profound atrophy in arm and fingers.
* Participants with severe cognitive dysfunction that would interfere with understanding instructions from the physician or therapist.
* Presence of any other musculoskeletal condition. e.g. (Frozen shoulder, any recent fractures of upper limb.
* Any accompanying diseases or disorders, other than stroke, that could interfere with upper extremity training.
* Uncontrolled health conditions for which exercise was contraindicated.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
1. Motor Evaluation Scale For Upper Extremity In Stroke Patients (MESUPES) | 8 week
  A 17-items into two sub scales ; MESUPES Arm function; 8 items(score 0-5) MESUPES-Hand function; 9 items (score0-2) objective evaluation scale designed to assess quality of movement of arm and hand function after stroke. MESUPES takes 5-15 min to complete. Total score 58. A higher score indicates the greater the quality of movement
2. Fugl-Meyer Assessment (FMA): | 8 weeks
  The Fugl-Meyer Assessment is used to assess motor function. It is a well-designed, feasible and efficient clinical examination method that has been tested widely in the stroke population. A three-level ordinal scale (0, can perform no part of the test; 1, performs test partially; 2, performs test normally) is applied to each item. A total possible score for the upper extremity is 66. The higher the score, the better the performance.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Jabeen, MS-NMPT, Study Chair — Riphah International University
Locations (1):
- Dr. Faisal Masood Teaching Hospital, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGregor HR, Cashaback JGA, Gribble PL. Somatosensory perceptual training enhances motor learning by observing. J Neurophysiol. 2018 Dec 1;120(6):3017-3025. doi: 10.1152/jn.00313.2018. Epub 2018 Sep 19. PMID 30230990
- [Background] Soltani Kouhbanani S, Arabi SM, Zarenezhad S, Khosrorad R. The Effect of Perceptual-Motor Training on Executive Functions in Children with Non-Verbal Learning Disorder. Neuropsychiatr Dis Treat. 2020 May 5;16:1129-1137. doi: 10.2147/NDT.S252662. eCollection 2020. PMID 32440127
- [Background] Bergmann F, Gray R, Wachsmuth S, Honer O. Perceptual-Motor and Perceptual-Cognitive Skill Acquisition in Soccer: A Systematic Review on the Influence of Practice Design and Coaching Behavior. Front Psychol. 2021 Dec 2;12:772201. doi: 10.3389/fpsyg.2021.772201. eCollection 2021. PMID 34925173
- [Background] Platzer WS. Effect of perceptual motor training on gross-motor skill and self-concept of young children. Am J Occup Ther. 1976 Aug;30(7):422-8. PMID 941962
- [Background] Fujimoto K, Ueno M, Etoh S, Shimodozono M. Combined repetitive facilitative exercise under continuous neuromuscular electrical stimulation and task-oriented training for hemiplegic upper extremity during convalescent phase after stroke: before-and-after feasibility trial. Front Neurol. 2024 Feb 22;15:1356732. doi: 10.3389/fneur.2024.1356732. eCollection 2024. PMID 38456153
- [Background] Purton J, Sim J, Hunter SM. Stroke survivors' views on their priorities for upper-limb recovery and the availability of therapy services after stroke: a longitudinal, phenomenological study. Disabil Rehabil. 2023 Sep;45(19):3059-3069. doi: 10.1080/09638288.2022.2120097. Epub 2022 Sep 15. PMID 36111388
- [Background] Hokazono A, Etoh S, Jonoshita Y, Kawahira K, Shimodozono M. Combination therapy with repetitive facilitative exercise program and botulinum toxin type A to improve motor function for the upper-limb spastic paresis in chronic stroke: A randomized controlled trial. J Hand Ther. 2022 Oct-Dec;35(4):507-515. doi: 10.1016/j.jht.2021.01.005. Epub 2021 Jan 26. PMID 33820711